CLINICAL TRIAL: NCT00153634
Title: Standard vs. Biofilm Susceptibility Testing in CF
Brief Title: Standard vs. Biofilm Susceptibility Testing in Cystic Fibrosis (CF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BURNS03A0
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2007-11

CONDITIONS: Cystic Fibrosis; Chronic Bronchitis
Keywords: Cystic fibrosis; Antibiotic susceptibility testing; Pseudomonas aeruginosa; Chronic bronchitis; Biofilms
MeSH Terms: conditions — Cystic Fibrosis; Bronchitis, Chronic; Pseudomonas Infections | interventions — Amikacin; Ceftazidime; Meropenem; Piperacillin, Tazobactam Drug Combination; ticarcillin-clavulanic acid; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Antibiotic regimen assignment based on biofilm susceptibility test results
  Interventions: Drug: IV amikacin; Drug: PO azithromycin; Drug: IV ceftazidime; Drug: PO ciprofloxacin; Drug: IV meropenem; Drug: IV piperacillin-tazobactam; Drug: IV ticarcillin-clavulanate; Drug: IV tobramycin
- 2 (Active Comparator): Antibiotic regimen assignment based on conventional susceptibility test results
  Interventions: Drug: IV amikacin; Drug: PO azithromycin; Drug: IV ceftazidime; Drug: PO ciprofloxacin; Drug: IV meropenem; Drug: IV piperacillin-tazobactam; Drug: IV ticarcillin-clavulanate; Drug: IV tobramycin

INTERVENTIONS:
Drug: IV amikacin — 5-7.5 mg/kg every 8 hrs or previous dose; start at previous recent stable dose then monitor serum levels and adjust dose, if needed, per standard clinical practice at the site
Drug: PO azithromycin — 250 mg once daily
Drug: IV ceftazidime — 50 mg/kg every 8 hours, up to 2 grams every 8 hours
Drug: PO ciprofloxacin — 500 mg every 12 hours if weight <50 kg 750 mg every 12 hours if weight ≥50 kg
Drug: IV meropenem — 40 mg/kg every 8 hours, up to 2 grams every 8 hours
Drug: IV piperacillin-tazobactam — 100 mg/kg of piperacillin component every 6 hours, up to 3 grams every 6 hours; antibiotic combination formulated in a fixed ratio, thus dosing is described for first component only
Drug: IV ticarcillin-clavulanate — 100 mg/kg of ticarcillin component every 6 hours, up to 3 grams every 6 hours; antibiotic combination formulated in a fixed ratio, thus dosing is described for first component only
Drug: IV tobramycin — 2.5-3.3 mg/kg every 8 hrs or previous dose; start at previous recent stable dose then monitor serum levels and adjust dose, if needed, per standard clinical practice at the site

SUMMARY:
This was a randomized multi-center clinical trial to compare the microbiological efficacy, clinical efficacy, and safety of using standard versus biofilm susceptibility testing of P. aeruginosa sputum isolates to guide antibiotic selection for treatment of airway infection in clinically stable patients with CF.

DETAILED DESCRIPTION:
Patients were screened to determine eligibility and to obtain a sputum culture. Eligible patients were randomized to either the standard or biofilm study arm. Antibiotic selection was performed centrally according to a standard algorithm using the susceptibility test results of the assigned study arm. On Day 0, patients were started on a 14-day course of two antibiotics as selected per protocol. Antibiotics were administered intravenously (IV) and/or orally. A follow-up phone call or visit occurred on Day 7. An end of treatment visit was conducted after completion of antibiotic therapy. A total of 39 patients were randomized. Many screened patients were ineligible for randomization based on microbiology results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on the following: sweat chloride > 60 mEq/L (by quantitative pilocarpine iontophoresis), or genotype with 2 identifiable mutations consistent with CF; and one or more clinical features consistent with CF.
* Age ≥ 14 years (changed from ≥ 18 years by protocol amendment).
* Able to expectorate sputum at screening.
* History of persistent positivity for P. aeruginosa on respiratory culture (at least three positive oropharyngeal (OP), sputum and/or bronchoscopy cultures in the 24 months prior to screening).
* Able to reproducibly perform pulmonary function testing.
* Clinically stable at screening, with no evidence of pulmonary exacerbation.
* Written informed consent provided.

Exclusion Criteria:

* Sputum culture negative for P. aeruginosa or density less than 10E5 CFU/gm at screening.
* Sputum culture positive for B. cepacia at screening.
* Presence of P. aeruginosa in sputum with off-scale resistance to all antibiotics by either method of susceptibility testing at screening. (changed from multiply-resistant P. aeruginosa by protocol amendment)
* History of B. cepacia positive respiratory culture within 24 months prior to screening.
* Hospitalization or treatment for a pulmonary exacerbation within 2 months prior to screening.
* Administration of parenteral anti-pseudomonal antibiotics within 2 months prior to screening.
* Treatment with oral or inhaled anti-pseudomonal antibiotics, or azithromycin or other macrolides within 14 days prior to screening.
* History of allergy (urticarial rash, diffuse erythroderma, serum sickness) to more than two groups of antibiotics (aminoglycosides, penicillins, cephalosporins, monobactams, macrolides, or quinolones) that are a therapeutic option.
* History of anaphylaxis or other life threatening complication to any antibiotic in the six groups that are a therapeutic option.
* History of abnormal renal function (serum creatinine > 1.5 x upper limit of normal) within one year of enrollment.
* History of abnormal liver function tests (> 2.5 x upper limit of normal) within one year of enrollment.
* Clinically documented hearing loss that precludes treatment with aminoglycosides.
* Post lung transplantation.
* Positive pregnancy test or female who is lactating or is not practicing an acceptable method of birth control.
* Presence of a condition or abnormality that in the opinion of an investigator would compromise the safety of the patient or the quality of the data.
* Administration of any investigational agent within 30 days prior to screening.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Microbiological efficacy: Change in P. aeruginosa density | from enrollment (up to day -21) to end of treatment (day 12-14)

SECONDARY OUTCOMES:
Clinical efficacy: Pre- to post-treatment change in FEV1 | from initiation (day 0) to end of treatment (day 12-14)
Safety: Adverse events, including new onset of acute pulmonary exacerbation and/or the need to change antibiotic therapy during the treatment period | from enrollment (up to day -21) to end of treatment (day 12-14)
Feasibility: Average costs and time per assay; rate of patient withdrawal because resistance patterns preclude randomization; self-reported technician satisfaction | during active enrollment (March 2004-November 2007)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Moskowitz, MD, Principal Investigator — Seattle Children's Hospital; Jane L Burns, MD, Study Chair — Children's Hospital and Regional Medical Center
Locations (8):
- United States (8):
  - University of Iowa, Iowa City, Iowa
  - Washington University St. Louis, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Background] Moskowitz SM, Foster JM, Emerson J, Burns JL. Clinically feasible biofilm susceptibility assay for isolates of Pseudomonas aeruginosa from patients with cystic fibrosis. J Clin Microbiol. 2004 May;42(5):1915-22. doi: 10.1128/JCM.42.5.1915-1922.2004. PMID 15131149
- [Background] Moskowitz SM, Foster JM, Emerson JC, Gibson RL, Burns JL. Use of Pseudomonas biofilm susceptibilities to assign simulated antibiotic regimens for cystic fibrosis airway infection. J Antimicrob Chemother. 2005 Nov;56(5):879-86. doi: 10.1093/jac/dki338. Epub 2005 Sep 27. PMID 16188918